CLINICAL TRIAL: NCT03747367
Title: The Microbiome and Responsiveness to Stress: Countermeasure Strategies for Improving Resilience to Sleep and Circadian Disruption (Experiments 1 & 2)
Brief Title: The Microbiome and Resilience to Sleep and Circadian Disruption
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Boulder (Other)
Collaborators: University of California, San Diego (Other); Office of Naval Research (ONR) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kenneth Wright, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15-0282
Record Dates: First submitted 2017-11-14; First posted 2018-11-20 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Sleep Deprivation; Circadian Dysregulation; Stress
Keywords: Microbiome; Stress; Sleep; Circadian
MeSH Terms: conditions — Sleep Deprivation; Chronobiology Disorders

STUDY DESIGN:
Intervention Model Description: Experiment 1 - Single group, repeated assessment Experiment 2 - Double-blind, randomized, cross-over design
Who Masked: Participant, Investigator
Masking Description: Experiment 1 - none Experiment 2 - double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): 8 hour sleep opportunity at habitual sleep/wake times for 14 days at home and 1 day in lab. Repeated for visit 1 and visit 2.
- Insufficient Sleep (Experimental): 3 days with 3 hour sleep opportunities in lab, immediately following baseline on both visit 1 and visit 2.
  Interventions: Behavioral: Insufficient Sleep

INTERVENTIONS:
Behavioral: Insufficient Sleep
  Arms: Insufficient Sleep

SUMMARY:
This study is about how sleep loss and being awake at night impacts the ability to think, changes molecules in the blood, and alters the bacteria that live in the gut that typically help keep people healthy. This work will have important implications for the development of treatments and countermeasures for people who do not sleep enough and need to be active at different times of the day and night (e.g., emergency workers and military personnel).

DETAILED DESCRIPTION:
Experiment 1: Consistency of microbiota-gut-brain axis responses

Prior to the start of this study, there are screening procedures to ensure participants meet the criteria for the study. At the first consent screening appointment, participants will learn more about the study, answer questionnaires, and complete a psychological interview. At the second medical screening appointment, participants will have a physical exam, blood work, drug screen, pregnancy test, electrocardiogram (a measurement of heart activity), and a resting metabolic rate assessment (a measurement of how much energy the body uses at rest). Participants will also meet with a nutritionist to discuss their food preferences for the study. Although participants are not financially compensated for the screening procedures, the expense of the screening tests is covered and copies are provided to the participant upon request. All of the results of the screening procedures are confidential and will only be used by the study staff to determine eligibility for the study.

Following the screening procedures, participants will complete two laboratory visits, both visits preceded by two weeks of home activity monitoring. During the home monitoring, participants wear a special watch that records activity levels. Participants also keep a sleep/wake log and use a website to log their daily sleep/wake times (if participants cannot access this website, they can call into an answering machine to inform investigators when they go to bed and wake up each day). The investigators will provide participants with a pre-study diet prepared by study dieticians for participants to eat for the three days prior to the laboratory visit. During the two weeks between the first and second laboratory visit participants will continue to wear the special watch, keep a sleep/wake log, and use a website to log their daily sleep/wake times (or call them into the answering machine). Participants will again be given a pre-study diet for the three days prior to their second visit.

During the laboratory visits, participants will live in the Sleep and Chronobiology Lab at the University of Colorado at Boulder for 3.7 days on two different occasions. The day before the inpatient visit begins, participants will spend the night in the laboratory, sleeping their normal 8 hours. This will be used as a pre-study screening for problems with sleep. In the morning participants will complete some pre-study tests and samples which will take approximately 60 minutes. Participants will then be permitted to leave the laboratory and in the evening they will return to begin the study. During the study participants sleep schedule will be changed to simulate the sleep loss that emergency workers in medical and military situations experience. Participants will be given an initial 3 hour sleep opportunity and then kept awake overnight. Throughout the study participants will be given a 3 hour sleep opportunity for every 24 hours of the laboratory visit. While participants are awake, they will be asked to perform a number of computer tasks, including a driving simulator. Blood and saliva samples will be taken to test for circadian and metabolic markers. Participants will also be asked to collect samples of the bacteria that live in their gastrointestinal tract from used bathroom tissue after they use the bathroom in the study. Finally, investigators will test how the heart and nervous system respond to stress by having participants place their hand in an ice water bath. At the end of the laboratory visit participants will be given an 11 hour sleep opportunity to recover from their sleep loss. After 3 more days of recovery sleep and another 2 weeks of home monitoring (identical to the first two weeks of the study), these procedures will be repeated in a second laboratory visit.

Experiment 2: Pre-biotic

Methods for experiment 2 are exactly the same as experiment 1 with the following addition: During the two weeks prior to laboratory visits, half of the study participants will be randomized (e.g., flip of a coin) to receive the prebiotic combination of polydextrose (PDX) and galacto-oligosaccharides (GOS) daily for 2 weeks and then tested in the first in-laboratory visit. These participants will then receive a maltodextrin placebo (a starch-derived food additive commonly used as a filling agent in a range of commercial foods and beverages) the two weeks prior to the second in-laboratory visit. The other half of participants will first receive maltodextrin and then the prebiotic diet. Investigators will provide participants the prebiotics and maltodextrin powders to be mixed in water and consumed each morning. The order in which participants receive the prebiotic diet will be maintained by the Clinical and Translational Research Center pharmacist. Neither the investigators nor participants will know what is in the powder provided.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Currently residing at Denver altitude or higher

Exclusion Criteria:

* Current major medical disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-10-21 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in fecal microbiome | Daily fecal samples while living in laboratory (3 samples per visit, 2 laboratory visits as part of a 39 day protocol)
  Fecal "beta diversity" (unit=weighted UniFrac)
Change in fecal metabolome | Daily fecal samples while living in laboratory (3 samples per visit, 2 laboratory visits as part of a 39 day protocol)
  Fecal small molecules (Mass spect metabolite abundance)

SECONDARY OUTCOMES:
Visual Search Performance | Assessed every 3 hours daily while living in the laboratory (17 times per visit, 2 laboratory visits as part of a 39 day protocol)
  Cognitive Throughput (items/minute)
Maintenance of wakefulness test | Assessed every 3 hours daily while living in the laboratory (17 times per visit, 2 laboratory visits as part of a 39 day protocol)
  Average latency to falling asleep (minutes)
Karolinska Sleepiness Scale | Assessed every 3 hours daily while living in the laboratory (17 times per visit, 2 laboratory visits as part of a 39 day protocol)
  Single question likert scale: Total score reported with a range of 1-9; min score=1[very alert], maximum score=9[very sleepy, great effort to keep awake, fighting sleep]. A higher score representing higher sleepiness. A lower score represents less sleepiness and a better outcome.
Changes in plasma metabolome | Assessed ~every 6 hours while living in the laboratory (10 times per visit, 2 laboratory visits as part of a 39 day protocol)
  Plasma small molecules (Mass spect metabolite abundance)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wright, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Sleep and Chronobiology Laboratory, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data generated from the proposed work that is presented in a peer reviewed journal will be de-identified.
  Microbiome data will be deposited in the International Nucleotide Sequence Database Collaboration www.insdc.org/ and is already deposited in Qiita http://qiita.microbio.me
  Metabolomics data will be deposited in Global Natural Products Social (GNPS) molecular networking http://gnps.ucsd.edu
  Other data that is presented in a peer reviewed journal will be archived indefinitely and made available upon request.
Time Frame: Upon publication, microbiome data to be deposited permanently in International Nucleotide Sequence Database Collaboration www.insdc.org/ Data already deposited in Qiita http://qiita.microbio.me Upon publication, metabolomics data to be deposited permanently in Global Natural Products Social (GNPS) molecular networking http://gnps.ucsd.edu
Access Criteria: data will be freely available at www.insdc.org/ and http://gnps.ucsd.edu